CLINICAL TRIAL: NCT02853968
Title: Unlock the Cell: Intracellular Inflammatory Pathways and Flow Cytometry Study for Castleman's Disease
Brief Title: Unlock the Cell: Castleman's Disease Flow Cytometry Study
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: Castleman Disease Collaborative Network (Other)
Responsible Party: Sponsor
Other Study IDs: 823546
Record Dates: First submitted 2016-07-15; First posted 2016-08-03 (Estimated); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Castleman Disease; Angiofollicular Lymphoid Hyperplasia; GLNH; Hyperplasia; Castleman's Disease; Angiofollicular Lymph Hyperplasia; Giant Lymph Node Hyperplasia
Keywords: Unlock the Cell; Castleman's Disease; CD; Castleman Disease; MCD; iMCD; Angiofollicular Lymph Hyperplasia; multicentric Castleman's disease; multicentric Castleman disease; idiopathic multicentric Castleman disease
MeSH Terms: conditions — Castleman Disease; Hyperplasia; Macular dystrophy, corneal type 1; Multi-centric Castleman's Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Our primary aim is to generate data to help to understand MCD pathogenesis, specifically: 1) what cells secrete cytokines, 2) what signaling pathways are activated, 3) what cytokines are released, and 4) what triggers this upregulation resulting in acute inflammation. We will investigate these samples using biochemical and RT-PCR techniques, proteomics, genomics, immunohistochemistry, storage for future use, cell culture treated with external stimuli, flow cytometry, and other molecular tests. We also want to collect excess stored tissue samples from previous procedures and store these samples along with unused blood samples and/or buccal swabs or saliva for future research purposes.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Castleman's Patients: Castleman's patients with HHV8 negative multicentric MCD
  Interventions: Procedure: Blood draw/buccal swab
- Related Disease Controls: Controls with inflammatory diseases similar to idiopathic multicentric Castleman's: i.e. HHV8+ MCD, HLH, Hodgkin disease
  Interventions: Procedure: Blood draw/buccal swab
- Healthy Donor Controls: Healthy subjects used for controls. These healthy subjects have no history of autoimmune disorders.
  Interventions: Procedure: Blood draw/buccal swab

INTERVENTIONS:
Procedure: Blood draw/buccal swab — The research project will need a blood sample of no more than 50mL per two month period. The research project may also request a buccal swab from patients if needed.

SUMMARY:
Castleman disease, a rare lymphoproliferative disorder, is characterized by inflammatory cytokine production and multiple organ system dysfunction. In this study, we will investigate inflammatory markers, cells, and signaling pathways in prospectively collected blood samples and/or buccal swabs or saliva using biochemical and RT-PCR techniques, proteomics, genomics, immunohistochemistry, storage for future use, cell culture treated with external stimuli, flow cytometry, and other molecular tests

DETAILED DESCRIPTION:
This is a University of Pennsylvania-sponsored project that is supported by the Castleman Disease Collaborative Network and the patients/loved one's group Castleman's Warriors (Castleman's Awareness and Research Effort).

Castleman Disease (CD) is a rare and poorly understood lymphoproliferative disease. The multicentric CD subtype (MCD) involves enlarged lymph nodes in multiple regions of the body and can be fatal if untreated. MCD patients demonstrate acute inflammatory crisis due to upregulation of inflammatory agents most notably IL-6 and VEGF followed by multiple organ failure and death.

Unlock the Cell aims to identify the pathways the disease takes through flow cytometry studies. The purpose of the CD Research study is to collect blood samples and/or buccal swabs or saliva samples and medical information of MCD patients and compare them to control samples so researchers can understand the causes of MCD, and design treatments based on our findings.

In this study, the investigators will analyze inflammatory markers, cells, and signaling pathways in prospectively collected blood samples using biochemical and RT-PCR techniques, proteomics, genomics, immunohistochemistry, storage for future use, cell culture treated with external stimuli, flow cytometry, and other molecular tests. A secondary aim is to collect excess stored tissue samples (e.g., lymph node, bone marrow) from previous procedures and store these samples along with unused blood samples for future research purposes to be performed at the University of Pennsylvania or shared with other Castleman disease researchers and biobanks.

ELIGIBILITY:
Inclusion Criteria:

* CD patients: Individuals of any age who are diagnosed with or suspected by a physician to have CD, including those who do have the ability to consent and those who lack the ability to consent
* Related Disease: Individuals who state that they have a disease that is a "Related Disease". "Related Disease" means autoimmune, oncology, inflammatory/lymphoproliferative disorders and infectious diseases that are similar to Castleman
* Healthy Individuals: Individuals without a history of auto-immune, inflammatory, infectious disease or oncologic disorders.

Exclusion Criteria:

• All individuals whose medical or psychological conditions (such as a mental handicap) would, in the opinion of the Principal Investigator, compromise the subject's safety or successful participation in the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals of any age (including those younger than 7 years of age), gender and ethnicity who have been diagnosed with CD
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
Collect PBMCs to use for inflammatory cell profiling via FACS | 1 year ~
  Peripheral blood will be collected to isolate peripheral blood mononuclear cells (PBMCs) used to look at inflammatory cell profiling via FACS. This will tell us what specific profiles are dysregulated.
Collect PBMCs to use for cell culture experiments | 1 year ~
  Peripheral blood will be collected to isolate peripheral blood mononuclear cells (PBMCs) for cell culture experiments.

SECONDARY OUTCOMES:
Use peripheral blood for biochemical testing | 1 year ~
  Biochemical testing will be performed on blood samples to collect inflammatory gene expressions using qPCR, ELISA and immunoblot.
Extract DNA and RNA from tissue samples to store in biobank | 1 year ~
  Excess blood sample tubes and/or buccal swabs or saliva will have DNA and RNA extracted and serum and plasma separated out to be stored in our biobank for future research.

CONTACTS AND LOCATIONS:
Overall Officials: Vera Krymskaya, PhD, MBA, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified Researchers, who apply for access to the data and are subsequently approved, will be given access to a limited dataset with direct identifiers removed in an Excel compatible file format or single SAS data files.
Supporting Information: Study Protocol, ICF

REFERENCES:
- See also: Hunt I: Columbia Hunt Pathogen Study — https://journals.plos.org/plosone/article?id=10.1371/journal.pone.0218660
- See also: Effectiveness of rituximab-containing treatment regimens in iMCD — https://www.ncbi.nlm.nih.gov/pubmed/29732477
- See also: iMCD International Treatment Guidelines — https://www.ncbi.nlm.nih.gov/pubmed/30181172

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-04-10): https://cdn.clinicaltrials.gov/large-docs/68/NCT02853968/Prot_SAP_ICF_000.pdf